CLINICAL TRIAL: NCT00053989
Title: Non-Myeloablative Allogeneic Hematopoietic Peripheral Blood Stem Cell Transplantation for Hematologic Malignancies and Disorders
Brief Title: NMA Allogeneic Hematopoietic Cell Transplant in Hematologic Cancer/Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269673; RP01-05
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-12

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Fanconi Anemia; Aplastic Anemia
Keywords: accelerated phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; primary myelofibrosis; de novo myelodysplastic syndromes; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; refractory anemia with excess blasts; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; Waldenstrom macroglobulinemia; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; adult acute myeloid leukemia in remission; secondary acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; childhood acute lymphoblastic leukemia in remission; adult acute lymphoblastic leukemia in remission; noncontiguous stage II adult lymphoblastic lymphoma; refractory multiple myeloma; refractory anemia; refractory chronic lymphocytic leukemia; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; grade 1 follicular lymphoma; grade 2 follicular lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Fanconi Anemia; Anemia, Aplastic; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelomonocytic, Chronic; Primary Myelofibrosis; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory, with Excess of Blasts; Waldenstrom Macroglobulinemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Hodgkin Disease; Leukemia, Myeloid, Acute; Anemia, Refractory; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Recurrence; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Antilymphocyte Serum; sargramostim; Cyclophosphamide; fludarabine phosphate; Methylprednisolone; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All patients enrolled on study
  Interventions: Biological: anti-thymocyte globulin; Biological: graft-versus-tumor induction therapy; Biological: sargramostim; Biological: therapeutic allogeneic lymphocytes; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methylprednisolone; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: allogeneic bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Procedure: umbilical cord blood transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin — iv
Biological: graft-versus-tumor induction therapy — iv
Biological: sargramostim — iv
Biological: therapeutic allogeneic lymphocytes — iv
Drug: cyclophosphamide — injection
Drug: fludarabine phosphate — iv
  Other Names: FLUDARA
Drug: methylprednisolone — oral
Drug: mycophenolate mofetil — oral
Drug: tacrolimus — oral
Procedure: allogeneic bone marrow transplantation — iv
Procedure: peripheral blood stem cell transplantation — iv
Procedure: umbilical cord blood transplantation — iv

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving immunosuppressive therapy before or after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well chemotherapy followed by donor peripheral stem cell transplant works in treating patients with hematologic cancer or aplastic anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxic effects of nonmyeloablative allogeneic peripheral blood stem cell transplantation in patients with a hematologic malignancy or aplastic anemia.
* Determine clinical response and overall outcome of patients treated with this regimen.
* Determine the incidence of graft-vs-tumor effect, graft-vs-host disease, and chimerism in patients treated with this regimen.

OUTLINE:

* Preparative regimen:

  * Matched related and unrelated donor transplantation:

    * Patients receive cyclophosphamide IV over 2 hours on days -5 and -4 and fludarabine IV over 30 minutes on days -5 to -1.
  * Cord blood transplantation:

    * Patients receive the same regimen as above plus anti-thymocyte globulin IV over 4 hours on days -3 to -1.
* Graft-vs-host disease (GVHD) prophylaxis:

  * Matched related and unrelated donor transplantation:

    * Patients receive oral tacrolimus (or IV) once daily and oral mycophenolate mofetil (MMF) (or IV) twice daily on days -1 to 60 followed by tapering* of this regimen. Patients then receive methotrexate IV on days 1, 3, and 6.
  * Cord blood transplantation:

    * Patients receive tacrolimus and MMF in the same regimen as above plus methylprednisolone twice daily on days 1-19 or until blood counts recover.
* Allogeneic stem cell reinfusion: Patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on day 0. Patients then receive sargramostim (GM-CSF) subcutaneously daily beginning on day 7 and continuing until blood counts recover.
* Donor lymphocyte infusion (DLI): Patients not converting to 100% donor T-cell chimerism by day 120 and showing signs of progresson of disease after tacrolimus and MMF withdrawal may receive DLI every 8 weeks for up to 3 infusions. Cord blood recipients do not receive DLI.

Patients are followed at day 100-120, every 3 months for 2 years, and then every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 30-60 patients will be accrued for this study within 6-7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of aplastic anemia

  * Severe disease
  * Failed at least 1 course of standard immunosuppressive regimen with cyclosporine and anti-thymocyte globulin OR
* Histologically confirmed hematologic malignancy including the following:

  * Acute leukemia

    * Any of the following types:

      * Acute myeloid leukemia (AML) with antecedent myelodysplastic syndromes
      * Secondary AML
      * AML with high-risk cytogenetic abnormalities
      * Acute lymphoblastic leukemia with high-risk cytogenetic abnormalities
    * Resistant or recurrent disease after combination chemotherapy with at least 1 standard regimen OR
    * In first remission at high risk of relapse
  * Chronic myelogenous leukemia

    * Chronic phase meeting at least 1 of the following criteria:

      * Failed imatinib mesylate
      * Failed interferon after at least 6 months of treatment with minimum of 21 million units of interferon per week
      * Unable to tolerate interferon
    * Accelerated phase (blasts less than 20%)
  * Myeloproliferative and myelodysplastic syndromes

    * Myelofibrosis (after splenectomy)
    * Refractory anemia
    * Refractory anemia with excess blasts
    * Chronic myelomonocytic leukemia
  * Lymphoproliferative disease

    * Chronic lymphocytic leukemia

      * Symptomatic disease after first-line chemotherapy
    * Low-grade non-Hodgkin's lymphoma (recurrent or persistent)

      * Symptomatic disease after first-line chemotherapy
    * Multiple myeloma

      * Progressive disease after autologous stem cell transplantation
    * Waldenstrom's macroglobulinemia

      * Failed 1 standard regimen
  * Non-Hodgkin's lymphoma meeting the following criteria:

    * Intermediate or high grade
    * Controlled and chemosensitive disease
    * First remission lymphoblastic or small non-cleaved cell lymphoma at high risk of relapse
  * Hodgkin's lymphoma

    * Relapsed and chemosensitive disease
* Not eligible for standard myeloablative allogeneic stem cell transplantation
* Availability of any of the following donor types:

  * Related donor matched at 5 or 6 HLA antigens (A, B, DR)
  * Unrelated donor fully matched by molecular analysis at A, B, DRB1, and DQB1 loci

    * Single antigen mismatch at C allowed
  * Cord blood that is 4, 5, or 6 match with recipient HLA antigens (A, B, DR) NOTE: No syngeneic donors permitted
* No uncontrolled CNS disease (for hematologic malignancies) NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 4 to 75 (if related or unrelated donor peripheral blood or marrow transplantation)
* 4 to 60 (if unrelated cord blood transplantation)

Performance status

* Karnofsky > 50%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin less than 3 times normal
* Alkaline phosphatase less than 3 times normal
* AST/ALT less than 3 times normal
* No Child's class B or C liver failure

Renal

* Creatinine clearance greater than 40 mL/min

Cardiovascular

* Cardiac ventricular ejection fraction at least 35% by MUGA
* No cardiovascular disease

Pulmonary

* DLCO at least 40% of predicted, corrected for hemoglobin and/or alveolar ventilation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV antibody negative
* No uncontrolled diabetes mellitus
* No active serious infection
* No other disease that would preclude study therapy
* No other concurrent malignancy except non-melanoma skin cancer
* No concurrent serious psychiatric illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* patients may have received a prior autologous blood or marrow transplantation (BMT)
* At least 6 months since prior allogeneic BMT

Chemotherapy

* See Disease Characteristics
* At least 2 weeks since prior chemotherapy, radiation or surgery

Endocrine therapy

* Not specified

Radiotherapy

* At least 2 weeks since prior radiotherapy

Surgery

* At least 2 weeks since prior surgery

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-01-29 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. McCarthy, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients enrolled on study Patients received cyclophosphamide 50 mg/kg on days -5 and -4, and fludarabine 25 mg/m2 on days -5, -4, -3, -2, -1.
  Hematopoietic cells from peripheral blood or marrow were infused on day 0. Patients who received hematopoietic cells from cord blood additionally received ATG 30 mg/kg on days -3, -2, -1.
  Fanconi anemia patients received cyclophosphamide 7.5 mg/kg on days -6, -5, -4, -3, fludarabine 25 mg/m2 on days -6, -5, -4, -3, -2 and ATG 30 mg/kg on days -3, -2, -1 and hematopoietic cells infused on day 0.
Period: Overall Study
Arm/Group | All Patients
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 37
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 52 [5 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41
Diagnosis [Count of Participants; unit: Participants]
  Acute lymphoblastic or myeloid leukemia | 12
  Hodgkin/non-Hodgkin lymphoma/prolymphocytic leukem | 21
  Multiple Myeloma | 2
  Myelodysplastic syndrome | 5
  Fanconi anemia | 1

OUTCOME MEASURES:

1. Primary Outcome: Day 100 TRM
Description: treatment related mortality within 100 days from hematopoietic stem cell (HSC) infusion on day 0
Time Frame: from start or conditioning (day -6 or -5) through day +100 after HSC infusion
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 41
Participants | 4

2. Primary Outcome: Day 100 Best Response
Description: Best disease response measured within 100 days from hematopoietic stem cell (HSC) infusion on day 0 using disease specific response criteria defined in the protocol
Time Frame: from start of conditioning on day -6 or -5 through day +100 after HSC infusion
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 41
Participants
  Complete Response | 22
  Partial Response | 5
  Early Death/NE | 4
  No Response/Stable Disease | 2
  Progressed | 8

3. Secondary Outcome: PFS
Description: Progression free survival defined as time from HSC infusion (day 0) until progression of disease or death due to any cause. Patients are censored if alive without disease progression through 1 year after HSC infusion
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 41
percentage of participants | 27 [13 to 40]

4. Secondary Outcome: OS
Description: Overall survival with events defined as death due to any cause and censored patients are alive as of 1 year post HSC infusion
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 41
percentage of participants | 44 [29 to 59]

5. Secondary Outcome: Acute GvHD
Description: overall grade II-IV acute GvHD
Time Frame: Day +100
Population: 2 participants died before they were eligible for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 39
Participants | 16

ADVERSE EVENTS:
Time Frame: 100 days
Description: SAE=died before absolute neutrophil count recovery (DBE) or survived to day +28 without absolute neutrophil count recovery (FTE) AE=overall grade III-IV acute GVHD
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 8/41
Serious Adverse Events (participants affected / at risk) | 3/41
Other Adverse Events (participants affected / at risk) | 6/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=41)
DBE/FTE (Blood and lymphatic system disorders) | 3 (3) — died before absolute neutrophil count recovery (DBE) or survived to day +28 without absolute neutrophil count recovery (FTE)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=41)
acute GVHD grade III-IV (Immune system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT00053989/Prot_SAP_000.pdf